CLINICAL TRIAL: NCT07084623
Title: Comparison of Pre-procedure Lignocaine Spray Versus Spray-as-you-go for Topical Airway Anesthesia in Flexible Bronchoscopy: A Randomized Controlled Trial
Brief Title: Comparison of Pre-procedure Lignocaine Spray Versus Spray-as-you-go for Topical Airway Anesthesia in Flexible Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Responsible Party: Principal Investigator, Talha Mahmud, Professor of Pulmonology, Sheikh Zayed Federal Postgraduate Medical Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SheikhZayedFederalPMER
Record Dates: First submitted 2025-06-04; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Lignocaine; Anesthesia, Local; Trachea; Airway Disease
MeSH Terms: conditions — Tracheal Diseases

STUDY DESIGN:
Intervention Model Description: A single-blind randomized controlled trial was conducted at the Pulmonology Department of Shaikh Zayed Hospital, Lahore, Pakistan, from March 2021 to March 2022.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-procedure lignocaine spray (PPL) (Active Comparator): Participants received:
  1. Standard sedation with midazolam (0.01 mg/kg IV);
  2. 2 mL of 4% lignocaine spray in the oropharynx before bronchoscopy;
  3. Additional 2% lignocaine spray (3 mg/kg):
     * 2-4 mL sprayed over vocal cords via bronchoscope working channel
     * Remaining dose as single bolus into larynx/trachea
  Interventions: Drug: Pre-procedure lignocaine spray (PPL); Drug: Lignocaine Spray (Spray-as-you-go)
- Spray-as-you-go (SAYG) Airway Anesthesia (Active Comparator): Participants received:
  1. Standard sedation with midazolam (0.01 mg/kg IV);
  2. 2 mL of 4% lignocaine spray in the oropharynx before bronchoscopy;
  3. 2% lignocaine spray (3 mg/kg) during procedure:
     * Initial 2-4 mL sprayed over vocal cords
     * Additional doses in mainstem bronchi during scope advancement
  Interventions: Drug: Pre-procedure lignocaine spray (PPL); Drug: Lignocaine Spray (Spray-as-you-go)

INTERVENTIONS:
Drug: Pre-procedure lignocaine spray (PPL) — Administration of 2 mL of 4% lignocaine spray in the oropharynx before the fiberoptic bronchoscopy procedure, followed by additional 2% lignocaine spray according to body weight (3 mg/kg)
Drug: Lignocaine Spray (Spray-as-you-go) — Administration of 2% lignocaine spray via oral scope insertion during the fiberoptic bronchoscopy procedure, according to body weight (3 mg/kg), with standard procedural sedation with midazolam and initial 2 mL of 4% lignocaine spray in the oropharynx for gag reflex suppression

SUMMARY:
Title: Comparing Two Methods of Topical Anesthesia for Fiberoptic Bronchoscopy

Purpose: To compare the effectiveness of two methods of anesthesia, pre-procedure lignocaine spray (PPL) and spray-as-you-go (SAYG), in reducing discomfort and improving operator comfort during fiberoptic bronchoscopy.

Study Design: Randomized controlled trial Participants: 50 patients undergoing fiberoptic bronchoscopy Interventions: Patients received either PPL or SAYG anesthesia

Outcomes:

* Pain perception
* Cough severity
* Operator comfort
* Procedure duration

Results:

* Both PPL and SAYG methods were effective in reducing pain and discomfort
* No significant differences were observed between the two groups in pain perception, cough scores, or procedure duration
* Operator comfort scores showed a trend favoring PPL, but the difference was not statistically significant

Implications: Both PPL and SAYG methods can be effectively used for fiberoptic bronchoscopy, with potential implications for procedural efficiency and patient outcomes.

DETAILED DESCRIPTION:
A single-blind RCT included 50 participants were randomly assigned to two groups (n = 25 each). Standard procedural sedation with midazolam and 2 mL of 4% lignocaine spray in the oropharynx was used to suppress the gag reflex. Additionally, 2% lignocaine spray was administered during the procedure according to body weight (3 mg/kg) via oral scope insertion. Cough severity, pain perception, and operator comfort were assessed using the Visual Analogue Scale, Faces Pain Rating Scale, and a 4-point Likert scale, respectively.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients indicated for diagnostic bronchoscopy, aged over 18 years, both genders (males and females), hemodynamically stable (defined as systolic blood pressure between 100 and 180 mm Hg), and sedated with an intravenous injection of midazolam at 0.01 mg/kg.

Exclusion Criteria:

* Hypersensitivity to lignocaine, use of general anesthesia for the procedure or other emergency procedures, pregnancy, comorbidities such as heart failure, advanced chronic kidney disease stage 3-4, chronic liver disease, contraindications to sedation, and hypoxemia (oxygen saturation by pulse oximetry, SpO2 < 92%)

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Patient discomfort and operator comfort during fiberoptic bronchoscopy | One year
  This composite outcome evaluates three distinct parameters:
  1. Cough severity measured by the Visual Analog Scale (100-mm scale where 0 mm indicates no cough and 100 mm indicates worst possible cough, with higher scores representing worse severity);
  2. Pain perception assessed via the Faces Pain Rating Scale (11-point scale from 0 [no pain] to 10 [worst imaginable pain], where higher scores indicate worse pain); and
  3. Operator comfort rated on a 4-point Likert scale (1 = Not comfortable to 4 = Very comfortable, with higher scores reflecting better comfort).
  All measures will be analyzed separately to compare PPL and SAYG techniques
Visual Analogue Scale | One year
  Cough severity measured using 100-mm Visual Analog Scale where 0 mm = no cough and 100 mm = worst cough imaginable. Higher scores indicate worse cough severity.
Faces Pain Rating Scale | One year
  Pain intensity measured using Faces Pain Rating Scale (0-10) where 0 = no pain and 10 = worst pain possible. Higher scores indicate worse pain.
4-point Likert scale | One year
  Operator comfort assessed via 4-point Likert scale where 1 = Not comfortable, 2 = Slightly uncomfortable, 3 = Comfortable, and 4 = Very comfortable. Higher scores indicate better comfort.

SECONDARY OUTCOMES:
Procedure duration | One year
  Comparison of procedure duration between PPL and SAYG airway anesthesia methods, measured in minutes from scope insertion to withdrawal.

OTHER OUTCOMES:
Comparative effectiveness of PPL versus SAYG anesthesia in cough suppression using the Visual Analog Scale (VAS) | One year
  This study will compare the effectiveness of pre-procedure lignocaine spray (PPL) and spray-as-you-go (SAYG) techniques in suppressing cough, measured by the Visual Analog Scale (VAS). The VAS is a 100-mm scale where 0 = no cough and 100 = worst cough, with higher scores indicating worse outcomes.
Comparative effectiveness of PPL versus SAYG anesthesia in pain control using the Faces Pain Rating Scale (FPRS) | One year
  This study will compare the effectiveness of PPL and SAYG techniques in pain control, assessed via the Faces Pain Rating Scale (FPRS). The FPRS is a 0-10 scale where 0 = no pain and 10 = worst pain, with higher scores indicating worse outcomes.
Comparative effectiveness of PPL versus SAYG anesthesia in operator comfort using the Operator Likert Scale | One year
  This study will compare the effectiveness of PPL and SAYG techniques in operator comfort, evaluated using a 4-point Likert scale (1 = Not comfortable, 4 = Very comfortable), with higher scores indicating better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Talha Mahmud, PhD, Principal Investigator — Shaikh Zayed Medical Complex, Federal Postgraduate Medical Institute, Lahore Pakistan.; Hira Ishtiaq, MD, Principal Investigator — Shaikh Zayed Medical Complex, Federal Postgraduate Medical Institute, Lahore Pakistan.
Locations (1):
- Shaikh Zayed Hospital, Federal Postgraduate Medical Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No